CLINICAL TRIAL: NCT05657639
Title: Venetoclax, Cladribine Plus Low-dose Cytarabine for Relapsed/Refractory Acute Myeloid Leukemia: a Multicenter, Randomized, Controlled Study
Brief Title: CAV Regimen for R/R AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: The Second People's Hospital of Huai'an (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Northern Jiangsu People's Hospital (Other); Affiliated Hospital of Nantong University (Other); Suzhou Hospital of Traditional Chinese Medicine (Other); Jining Medical University (Other); The First People's Hospital of Changzhou (Other); The First Affiliated Hospital of Anhui Medical University (Other); First Affiliated Hospital of Zhejiang University (Other); YANCHENG NO.1 PEOPLE'S HOSPITAL (Unknown); Kaifeng Central Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Professor, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZAML02
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: venetoclax; cladribine; cytarabine; relapsed/refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CAV regimen; MEC regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAV regimen (Experimental)
  Interventions: Drug: CAV Regimen
- MEC regimen (Active Comparator)
  Interventions: Drug: MEC Regimen

INTERVENTIONS:
Drug: CAV Regimen — Cladribine 5 mg/m2/day , cytarabine 20mg q12h, venetoclax 100mg d1, 200 d2, 400 mg/day from day 3 to day 21.
  Arms: CAV regimen
Drug: MEC Regimen — Mitoxantrone 8mg/m2 d1-5, etoposide 100mg/m2 d1-5, cytarabine 1g/m2 d1-5
  Arms: MEC regimen

SUMMARY:
This study aims to investigate the efficacy and safety of cladribine, combined with low-dose cytarabine and venetoclax (CAV regimen) for relapsed/refractory acute myeloid leukemia (R/R AML).

DETAILED DESCRIPTION:
Patients with relapse/refractory (R/R) acute myeloid leukemia often show resistance to conventional chemotherapy and have dismal prognosis. Salvage therapy using venetoclax combined with hypomethylation drugs achieved an overall response rate of only approximately 40% in R/R AML. Cladribine, a purine analogue, exerts cytotoxic, proapoptotic, and antiproliferative effects on AML cells.The efficacy of cladribine plus cytarabine and venetoclax in R/R AML has not been reported.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16-70 years old.
2. Diagnosed with R/R AML.
3. Patients with AML must meet one of the following criteria, A or B: A: Refractory AML disease was defined as follows: (1) failure to attain CR following exposure to at least 2 courses of standard or intensive induction therapy; or (2) bone marrow leukemia cell decline index (BMCDI) < 50% and > 20% after 1 course of standard or intensive induction therapy. B: Relapsed AML disease was defined as follows:

(1) reappearance of leukemic blasts in the peripheral blood after CR; or (2) detection of ≥ 5% blasts in the BM not attributable to another cause (e.g., BM regeneration after consolidation therapy); or (3) extramedullary relapse.

4. ECOG performance status score less than 2. 5. Expected survival time ≥12 weeks. 6. Without serious heart, lung, liver, or kidney dysfunction. 7. Able to understand and provide informed consent.

Exclusion Criteria:

1. Patients who are allergic to the study drug or drugs with similar chemical structures.
2. Pregnant or lactating women, and women of childbearing age who do not want to practice effective methods of contraception.
3. Active infection.
4. Active bleeding.
5. Patients with new thrombosis, embolism, cerebral hemorrhage, or other diseases or a medical history within one year before enrollment.
6. Patients with mental disorders or other conditions.
7. Liver function abnormalities (total bilirubin > 1.5 times of the upper limit of the normal range, ALT/AST > 2.5 times of the upper limit of the normal range or patients with liver involvement whose ALT/AST > 1.5 times the upper limit of the normal range), or renal dysfunction (Ccr<50ml/h).
8. Patients with a history of clinically significant QTc interval prolongation (male > 450 ms; female > 470 ms), ventricular heart tachycardia and atrial fibrillation, II-degree heart block, myocardial infarction attack within one year before enrollment, and congestive heart failure, and patients with coronary heart disease who have clinical symptoms and requiring drug treatment.
9. Patients who relapsed after allogeneic hematopoietic stem cell transplantation.
10. Drug abuse or long-term alcohol abuse that would affect the evaluation results.
11. Patients who have received organ transplants.
12. Patients not suitable for the study according to the investigator's assessment.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | ORR assessment is measured on days 21 from the start of CAV regimen
  The overall response (completed remission, completed remission with incomplete blood count recovery, morphologic leukemia-free state and partial remission)

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  OS is measured from the time of enrollment to this study to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Event-free survival (EFS) | 2 years
  EFS is measured from the time of enrollment to this study to treatment failure or relapse or any cause of death.
Treatment-related mortality (TRM) | 2 months
  Death due to treatment (within 8 weeks) during and after completion of chemotherapy.
Adverse events (AEs) | 2 months
  It is evaluated and graded according to CTCAE 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No